CLINICAL TRIAL: NCT01030055
Title: A Randomized, Open-label, Multi-center, Phase I, Crossover Study to Assess the Relative Bioavailability of 2 Oral Formulations of TKI258, and the Effect of Food on the Bioavailability of TKI258, in Patients With Advanced Solid Tumors
Brief Title: Bioavailability and Food Effect Study of TKI258 (CSF Capsules vs. FMI Capsules)in Adult Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CTKI258A2112
Record Dates: First submitted 2009-12-08; First posted 2009-12-11 (Estimated); Last update posted 2020-12-21 (Actual); Status verified 2013-12

CONDITIONS: Neoplasms; Cancer; Tumors
Keywords: Neoplasms; Cancer; Tumors; Administration, oral; Capsules; CHIR258; CHIR-258; CHIR 258; TKI258; TKI-258; TKI 258; Bioavailability; Food
MeSH Terms: conditions — Neoplasms | interventions — 4-amino-5-fluoro-3-(5-(4-methylpiperazin-1-yl)-1H-benzimidazol-2-yl)quinolin-2(1H)-one

ARMS (2):
- TKI258 - bioavailability (Experimental)
  Interventions: Drug: TKI258 (dovitinib)
- TKI258 - food (Experimental)
  Interventions: Drug: TKI258 (dovitinib)

INTERVENTIONS:
Drug: TKI258 (dovitinib) — bioavailability (anhydrate capsules) food (monohydrae capsules)
  Other Names: dovitinib

SUMMARY:
This study will evaluate the relative bioavailability of 2 oral formulations of TKI258, and the effect of food on the bioavailability of TKI258, in adult patients with advanced solid tumor

ELIGIBILITY:
Inclusion Criteria:

* Patients with an advanced solid tumor, except breast cancer,which has progressed despite standard therapy, or for which no standard therapy exists
* World Health Organization (WHO) performance status ≤ 2
* Patient must meet protocol-specified laboratory values

Exclusion Criteria:

* Patients with brain cancer
* Patients who have concurrent severe and/or uncontrolled medical conditions which could compromise participation in the study
* Patients who have not recovered from previous anti-cancer therapies
* Female patients who are pregnant, breast feeding, or not willing to use an effective method of birth control

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-02; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Determine the relative bioavailability of the final market image form of TKI258 (monohydrate capsules) as compared to the clinical service form of TKI258 (anhydrate capsules) | 9 days
Determine the effect of food on the bioavailability of TKI258 | 22 days

SECONDARY OUTCOMES:
Characterize the safety and tolerability of TKI258, including acute and chronic toxicities | Up to 28 days after the last dose of study drug
Evaluate preliminary evidence of anti-tumor activity of TKI258 in patients with advanced solid tumors. | Every 8 weeks until progression of disease

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (4):
- United States (4):
  - City of Hope National Medical Center, Duarte, California
  - University of California at Los Angeles, Los Angeles, California
  - Duke University Medical Center Cancer Dept, Durham, North Carolina
  - University of Utah / Huntsman Cancer Institute, Salt Lake City, Utah

REFERENCES:
- See also: Results for CTKI258A2112 can be found on the Novartis Clinical Trial Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=8983